CLINICAL TRIAL: NCT05531409
Title: Responsible Behavior With Younger Children (RBYC) Pilot Study
Brief Title: Responsible Behavior With Younger Children Pilot Study
Acronym: RBYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of Virginia (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00007351
Record Dates: First submitted 2022-06-28; First posted 2022-09-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2022-09

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Pilot randomized waitlist-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Students from 6th and 7th grades from two schools were randomized to receive the RBYC curriculum. The RBYC curriculum has eight core content sessions, each of which lasts approximately 45 minutes. These include sessions that address: 1) Developmental differences between children versus teenagers; 2) Perspective-taking of and empathic responding to younger children; 3) and 4) Healthy versus unhealthy teenage-younger child relationships; 5) Misconceptions versus facts about child sexual abuse and legal ramifications; 6) Why adolescents may engage in harmful sexual behaviors; 7) Peer sexual harassment, what it is and how to avoid or address it; and 8) Being a good bystander or upstander when you have concerns that another child or peer has been or may be harmed. The RBYC curriculum was integrated into each school's existing health education curriculum.
  Interventions: Behavioral: Responsible Behavior for Younger Children (RBYC)
- Waitlist Control (No Intervention): Students from 6th and 7th grades from the two schools that were randomized to the waitlist control condition received the RBYC curriculum once the study was completed (i.e., baseline and post-assessment data were collected).

INTERVENTIONS:
Behavioral: Responsible Behavior for Younger Children (RBYC) — RBYC is a school-based universal prevention program designed to provide adolescents and their parents (or other guardians) with the knowledge and tools to help adolescents interact appropriately with younger children and avoid engaging younger children in sexual behaviors.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study was to develop and pilot test a universal school-based prevention curriculum to prevent the onset of child sexual abuse (CSA) perpetration by early adolescents against younger children.

DETAILED DESCRIPTION:
The proposed Responsible Behavior with Younger Children (RBYC) curriculum was developed and pilot tested in 6th and 7th grade classes in Baltimore City Public Schools. This study had three aims: 1) to develop and refine a new classroom-based universal curriculum to prevent the onset of CSA perpetration, 2) to evaluate the immediate effects (pre-post design) of RBYC on targeted constructs, and 3) to determine the feasibility and acceptability of RBYC to youth, parents, and school personnel.

ELIGIBILITY:
Inclusion Criteria:

* Student Assessments: 1) are in a 6th or 7th grade class within one of the four participating schools, 2) are fluent in English, and 3) have a "yes" consent form completed by their parent/legal guardian; students will also be asked to complete an electronic assent form at the beginning of each of the three student assessments.
* Educator Interviews: 1) have witnessed at least one session of the RBYC curriculum, 2) are fluent in English, and 3) have completed a consent form

Exclusion Criteria:

* Children residing in foster care will not be eligible for participation because of challenges associated with obtaining written parental consent from the legal guardian and other clinical concerns regarding this potentially vulnerable population that may arise with either students or parents. It is not feasible to address these challenges in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Developmental Differences Between Children and Adolescents | 2 months
  RBYC aims to educate children about developmental differences between adolescents and younger children. The investigators were unable to identify an existing relevant measure and therefore created seven items to assess knowledge about developmental differences between adolescents and younger children. For example, "Children might feel frustrated when they can't do the same things as teenagers." Response options were true or false and scored as 0 (inaccurate) or 1 (accurate). Scale range = 0-7, with higher scores indicating more accurate understanding of developmental differences between teenagers and younger children.
Knowledge about CSA and Related Concepts | 2 months
  Included 41 true/false items coded as 0 (inaccurate) or 1 (accurate) to assess five core areas of knowledge reflecting five subscales: child sexual abuse facts, child sexual abuse laws, child sexual abuse prevention, knowledge about sexual harassment, knowledge about sexual consent Items comprising a given subscale were summed for a subscale score, with higher scores indicating more accurate knowledge.Items were created by the investigators for the study and also adapted from: Adolescent Cognition Scale (Hunter, Becker, Kaplan, & Goodwin, 1991), Children's Knowledge of Abuse Questionnaire (Tutty, 1995), and Questionnaire on Child Sexual Abuse (Halpérin et al., 1996).
Peer Sexual Harassment Behaviors | 2 months
  Included five items assessing peer sexual harassment perpetration created by Taylor and colleagues (2011). For example "Have you ever done any of the following with a peer: Made sexual comments, jokes, gestures, or looks to them?" Response options were no (0) or yes (1) and were summed to provide a final score that ranged from 0-5 with higher scores indicating engaging in more harassing behaviors.
Behavioral Intention to Avoid or Prevent Harm | 2 months
  To assess intention to avoid peer sexual harassment, the investigators used five items developed by Taylor and colleagues (Taylor et al., 2011). For example "I can help prevent sexual harassment against peers at my school". Items were measured on a four-point scale ranging from completely disagree (1) to completely agree (4) and summed for scores ranging from 5-20. To assess intention to avoid or prevent CSA, the investigators crafted seven similar items. For example "I know how to teach my friends about how to stop child sexual abuse". Again, response options ranged from completely disagree (1) to completely agree (4) and were summed for scores ranging from 7-28. For both scales, higher scores indicated stronger intention to prevent or avoid harm.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Letourneau, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health